CLINICAL TRIAL: NCT00388934
Title: Randomized Clinical Comparison of Cypher Select and Taxus Express Stent Implantation in Unselected Patients With Coronary Artery Disease.
Brief Title: Comparison of Cypher Select and Taxus Express Coronary Stents
Acronym: SORT-OUTII
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: University of Aarhus (Other); University of Copenhagen (Other); Odense University Hospital (Other)
Responsible Party: Department of Cardiology B, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SORT-OUT II
Record Dates: First submitted 2006-10-16; First posted 2006-10-17 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2007-05

CONDITIONS: Coronary Artery Disease; Angina Pectoris
Keywords: Percutaneous coronary intervention; Angina pectoris; Stent
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug eluting stent (Cypher) (Experimental): Percutaneous coronary intervention with implantation of drug eluting coronary stent (Cypher)
  Interventions: Device: Drug eluting stent
- Drug eluting stent (Taxus) (Experimental): Percutaneous coronary intervention with implantation of drug eluting coronary stent (Taxus)
  Interventions: Device: Drug eluting stent

INTERVENTIONS:
Device: Drug eluting stent — percutaneous intervention with implantation of drug eluting coronary stent
  Other Names: DES; Cypher; Taxus

SUMMARY:
Randomized nine months clinical comparison of implantation of Taxol eluting (Taxus Express) and Sirolimus eluting (Cypher Select) stents in non-selected patients with coronary artery disease.

DETAILED DESCRIPTION:
Design:

* Randomized open multicentre trial.

Patients:

* 1800 patients with coronary artery disease scheduled for percutaneous coronary intervention with stent implantation.

Inclusion criteria:

* Patients with coronary artery disease scheduled for percutaneous coronary intervention with stent implantation.
* Signed informed consent.

Exclusion criteria:

* Participation in other stent studies.

Randomization:

* Implantation of Taxus Express og Cypher Select stents.

Primary end-point:

* Combined end-point of cardiac death, new revascularization (PCI or CABG) or myocardial infarction after nine months.

Secondary end-points:

* Total death after nine months
* Cardiac death after nine months
* Myocardial infarction after nine months
* Index vessel myocardial infarction after nine months
* Target lesion revascularization
* Target vessel revascularization
* Stent thrombosis after nine months

End-point evaluation:

* End-points will be adjudicated by an independent end-point committee

ELIGIBILITY:
Inclusion Criteria:

* Planned implantation of drug eluting stent
* Written informed consent

Exclusion Criteria:

* Planned intervention with other stents than study stents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2095 (Actual)
Dates: Start 2004-08; Primary Completion 2006-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
MACE (cardiac death, myocardial infarction, target vessel revascularisation, target lesion revascularisation, TVF) | during 9 months

SECONDARY OUTCOMES:
Total death | after 9 months, 2 and 3 years
Cardiac death | after 9 months, 2 and 3 years
Myocardial infarction | after 9 months, 2 and 3 years
Target vessel revascularisation, target lesion revascularisation, TVF | after 9 months, 2 and 3 years
Stent thrombosis | after 9 months, 2 and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Anders Galloe, MD, Principal Investigator — Gentofte Hospital, Copenhagen

REFERENCES:
- [Derived] Galloe AM, Kelbaek H, Thuesen L, Hansen HS, Ravkilde J, Hansen PR, Christiansen EH, Abildgaard U, Stephansen G, Lassen JF, Engstrom T, Jensen JS, Jeppesen JL, Bligaard N; SORT OUT II Investigators. 10-Year Clinical Outcome After Randomization to Treatment by Sirolimus- or Paclitaxel-Eluting Coronary Stents. J Am Coll Cardiol. 2017 Feb 14;69(6):616-624. doi: 10.1016/j.jacc.2016.11.055. PMID 28183505
- [Derived] Galloe AM, Thuesen L, Kelbaek H, Thayssen P, Rasmussen K, Hansen PR, Bligaard N, Saunamaki K, Junker A, Aaroe J, Abildgaard U, Ravkilde J, Engstrom T, Jensen JS, Andersen HR, Botker HE, Galatius S, Kristensen SD, Madsen JK, Krusell LR, Abildstrom SZ, Stephansen GB, Lassen JF; SORT OUT II Investigators. Comparison of paclitaxel- and sirolimus-eluting stents in everyday clinical practice: the SORT OUT II randomized trial. JAMA. 2008 Jan 30;299(4):409-16. doi: 10.1001/jama.299.4.409. PMID 18230778